CLINICAL TRIAL: NCT03740126
Title: Surveillance With PET/CT and Liquid Biopsies of Stage I-III Lung Cancer Patients After Completion of Definitive Therapy; a Randomized Controlled Trial
Brief Title: Surveillance With PET/CT and Liquid Biopsies of Stage I-III Lung Cancer Patients After Completion of Definitive Therapy
Acronym: SUPE_R
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Lung Cancer Group (Other); Danish Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Barbara Malene Fischer, Senior Consultant, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-18009536
Record Dates: First submitted 2018-10-25; First posted 2018-11-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Positron Emission Tomography Computed Tomography; X-Ray Computed Tomography; Liquid Biopsy; Quality of Life; Medical Oncology; Radiation Oncology; Follow-up
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A, PET/CT (Experimental): 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography with computed tomography (FDG PET/CT) replacing computed tomography (CT) at months 6, 12, 18 and 24, otherwise as B with CT scan months 9, 15 and 21. Quality of life assessment and liquid biopsy every 3 months for later analysis.
  Interventions: Diagnostic Test: Whole body 18F-FDG PET/CT
- Control arm B (No Intervention): CT-scan and clinical evaluation every 3 months. Quality of life assessment and liquid biopsy at every 3 months for later analysis.

INTERVENTIONS:
Diagnostic Test: Whole body 18F-FDG PET/CT — In the experimental arm (A), an FDG-PET/CT scan will replace the CT-scan at 6, 12, 18 and 24 months post-treatment. A standard CT-scan will be performed at 3, 9, 15 and 21 months post-treatment. All patients will be asked for a blood sample for liquid biopsy and to fill in a quality of life questionnaire, concurrently every 3 months.
  Arms: Arm A, PET/CT

SUMMARY:
The purpose of this study is to improve early detection of treatable relapse of lung cancer and thereby improve survival and quality of life for the patients. The investigators will perform a multicenter, randomized controlled trial to 1) assess if surveillance with whole body Positron Emission Tomography combined with Computer Tomography (PET/CT) including the brain can increase the number of treatable relapses and 2) concurrently collect liquid biopsies for later analysis, potentially enabling even earlier and minimally invasive detection and characterization of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-small cell lung cancer (NSCLC), proven by cytology or histology
* Patient in clinical stages I-III
* Age≥ 18 years
* Performance status ≤ 2 at the time of referral to therapy
* Patient referred for definitive treatment (e.g. surgery, surgery followed by adjuvant chemotherapy, concomitant radio-chemotherapy, conventional or stereotactic radiotherapy or radiofrequency ablation).
* Patient has given his/her written informed consent before any specific procedure from protocol

Exclusion Criteria:

* Patient, whose disease has progressed within the first 3 months after cancer treatment, e.g. confirmed progressive disease on CT.
* Persons deprived of liberty or under guardianship or curators
* Dementia, mental alteration, severe psychiatric disease or other circumstances that can compromise informed consent from the patient and/or adherence to the protocol and the monitoring of the trial
* Pregnant or breastfeeding women
* Patient participating in another interventional study during the surveillance period. This is only relevant for studies that might interfere with the intervention, whereas studies on late effects will not preclude participation in SUPE-R. Participation in protocols related only to initial treatment will not preclude participation in SUPE-R. Cases of doubt will be settled by the steering committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of relapses treatable with curative intent | Until first detected relapse or 2 years after enrollment
  As decided by multidisciplinary meetings

SECONDARY OUTCOMES:
Time to verified relapse | From date of randomization until the date of first documented relapse assessed up to 24 months
  Relapse verified by histology or imaging combined with MDM review
Overall survival | From date of randomization until the date of censoring or death from any cause, whichever came first, assessed up to 36 months
  Death of any course or censoring
Overall survival for patients with relapse | From randomization until 12 months after first detected relapse or until death (whichever comes first)
  Death of any course or censoring
Performance status at relapse | From randomization until first detected relapse or 24 months
  Performance status of study participants at relapse will be assessed using Eastern Cooperative Oncology Group (ECOG) performance status scale from grade 0 to grade 4, where grade 0 corresponds to a patient who is "fully active, able to carry on all pre-disease performance without restriction" and grade 4 is a patient who is "completely disabled; cannot carry on any selfcare; totally confined to bed or chair".
Quality of life / QLQ-C30 | From randomization until first detected relapse or 24 months
  Quality of life will be assessed every 3rd month using a validated questionnaire, European Organisation for Research and Treatment of Cancer Quality of Life Questionaire Core Questionaire 30 (EORTC QLQ-C30).
  The questionaire is filled out by study participants at each control visit and patients score severity of a range of symptoms during the past week on a scale of 1 ("Not at all") to 4 ("Very much").
Quality of life / QLQ-LC13 | From randomization until first detected relapse or 24 months
  Quality of life will be assessed every 3rd month using a validated questionnaire, European Organisation for Research and Treatment of Cancer Quality of Life Questionair Lung Cancer 13 (EORTC QLQ-LC13).
  The questionaire is filled out by study participants at each control visit and patients score severity of a range of symptoms during the past week on a scale of 1 ("Not at all") to 4 ("Very much").
Quality of life / Raw score | From randomization until first detected relapse or 24 months
  From the results of QLQ-C30 and QLQ-LC13 a Raw Score (RS) is calculated (average of all scores) and Quality of Life is calculated as (RS - 1)/3 which outputs a value between 0 and 1, where 0 is a complete absence of symptoms and 1 is the maximum severity of all related symptoms. This will be used for calculation of QALY in the cost-effectiveness analysis.
Number of procedures to assess incidental findings | From randomization until 24 months or first detected relapse or until death (whichever comes first)
  Procedures resulting from an incidental finding on a follow up scan
Types of procedures to assess incidental findings | From randomization until 24 months or first detected relapse or until death (whichever comes first)
  Invasive / non-invasive
Adverse events due to invasive procedures done to assess incidental findings | From randomization until 24 months or first detected relapse or until death (whichever comes first)
  For example: Bleeding, pneumothorax, hospital admission
Cost-effectiveness analysis of intervention | From randomization until 24 months or 12 months after first detected relapse or until death (whichever comes first)
  Cost-effectiveness of the PET/CT regimen vs the CT regimen is assessed with the ICER (incremental cost-effectiveness ratio), i.e. the ratio of net health care costs to net QALYs ( quality-adjusted life years). Net health care costs are estimated as the health care costs difference between the two arms and net QALYs likewise. Health care costs are calculated from register-based information on health care consumption cumulated in 2-yrs follow-up (DRG-rates) supplemented by intervention costs based on project costs. The relevant cost data are available at "Sundhedsdatastyrelsen" using their research service.
Type of treatment after verification of relapse | From randomization until 12 months after first detected relapse or until death (whichever comes first)
  Description of treatment - e.g. surgical, radiotherapy, stereotactic ablative body radiotherapy, medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Fischer, MD PhD DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Gentofte Municipality
  - Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guldbrandsen KF, Bloch M, Skougaard K, Albrecht-Beste E, Nellemann HM, Krakauer M, Gortz PM, Gruner JM, Fledelius J, Nielsen AL, Holdgaard PC, Nielsen SS, Hjorthaug K, Ahlborn LB, Jakobsen E, Hojsgaard A, Petersen RH, Moller LB, Dahl M, Sorensen BS, Frank MS, Ehlers JH, Saghir Z, Pohl M, Borissova S, Land LH, Kristiansen C, McCulloch T, Mortensen LS, Christophersen MS, Hilberg O, Rasmussen TL, Schwaner SHS, Laursen CB, Bodtger U, Lonsdale MN, Meyer CN, Gerke O, Mortensen J, Rasmussen TR, Fischer BM; SUPE_R Study Group. Diagnostic Accuracy of [18F]FDG PET/CT versus CT for NSCLC Surveillance: Secondary Analysis of a Randomized Clinical Trial. Clin Lung Cancer. 2025 Nov 19:S1525-7304(25)00319-5. doi: 10.1016/j.cllc.2025.11.011. Online ahead of print. PMID 41387040
- [Derived] Guldbrandsen KF, Bloch M, Skougaard K, Ahlborn LB, Jakobsen E, Hojsgaard A, Petersen RH, Moller LB, Dahl M, Sorensen BS, Frank MS, Ehlers JH, Krakauer M, Gortz PM, Albrecht-Beste E, Gruner JM, Saghir Z, Fledelius J, Nielsen AL, Holdgaard PC, Nielsen SS, Pohl M, Borissova S, Land LH, Kristiansen C, McCulloch T, Mortensen LS, Nellemann HM, Christophersen MS, Hilberg O, Rasmussen TL, Schwaner SHS, Laursen CB, Bodtger U, Sopina L, Lonsdale MN, Meyer CN, Gerke O, Mortensen J, Rasmussen TR, Fischer BM; SUPE_R Study Group. Surveillance With Fluorine-18 Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography of Patients With Stage I-to-III Lung Cancer After Completion of Curative treatment (SUPE_R): A Randomized Controlled Trial. J Thorac Oncol. 2025 Aug;20(8):1086-1097. doi: 10.1016/j.jtho.2025.04.003. Epub 2025 Apr 19. PMID 40258572